CLINICAL TRIAL: NCT07196098
Title: Effect of Slow Tempo Music on Anxiety Markers During Intravitreal Injection: A Randomised Controlled Trial
Brief Title: Using Gentle Music to Ease Anxiety in People Receiving Eye Treatment Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ng Yu Siang (Other)
Responsible Party: Sponsor-Investigator, Ng Yu Siang, Doctor, University of Malaya
Organization: University of Malaya (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202424-13359
Record Dates: First submitted 2025-08-25; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Pain; Anxiety
Keywords: intravitreal injection; salivary alpha amylase; music intervention; anxiety; pain
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A repeated-measures, randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No background music was played before and during intravitreal injections
- Music Group (Experimental): Slow tempo music will be played 15 minutes before and during intravitreal injection.
  Interventions: Other: Slow tempo music

INTERVENTIONS:
Other: Slow tempo music — Slow tempo music will be played 15 minutes before and during intravitreal injection.
  Arms: Music Group

SUMMARY:
The goal of this clinical trial was to investigate the effects of slow tempo music on anxiety and perceived pain in patients undergoing elective intravitreal injections (IVI). The main questions it aimed to answer were:

Did slow tempo music reduce the anxiety and pain of patients undergoing IVI?

Did the pain threshold differ among patients of different ethnic groups?

Participants were divided into a music intervention group and a control group. Participants in the music group listened to slow tempo music before and during IVI, while participants in the control group received IVI without background music.

The study compared salivary alpha-amylase (sAA) levels-an enzyme that correlates with anxiety level-along with blood pressure (BP) and heart rate (HR) of participants before and after IVI. At the end of the treatment, participants' pain scores were obtained.

DETAILED DESCRIPTION:
Intravitreal injection (IVI) is a procedure in which medication is administered directly into the vitreous cavity. Since the introduction of anti-vascular endothelial growth factor (anti-VEGF) therapy two decades ago, the number of IVIs performed has increased substantially. These injections are now routinely conducted as outpatient procedures for the treatment of various retinal disorders such as diabetic macular edema (DME), age-related macular degeneration (AMD), retinal vein occlusion (RVO), polypoidal choroidal vasculopathy(PCV), and pseudophakic cystoid macular oedema.

Eligible participants were identified among patients scheduled for intravitreal injections (IVI) at the day-care surgery unit of the University of Malaya Medical Centre. Written informed consent was obtained after participants were provided with the participant information sheet and screened based on the study's inclusion and exclusion criteria. A simple random sampling method was used. After consent, each participant was randomly assigned a number using the Random Number Generator from the website https://www.calculatorsoup.com

, which generates numbers without repeats. Odd numbers were allocated to the music intervention group, and even numbers to the control group.

Data collection followed the Data Collection Proforma. Demographic information included age, gender, ethnicity, marital status, comorbid conditions, occupation, and education level. Before entering the operating room (OR), participants' baseline blood pressure (BP₀) and heart rate (HR₀) were recorded.

In this study, a standardised, copyright- and royalty-free piano composition-Andromeda (Piano Solo) by Gabriele Tosi, available for free on YouTube.com-was used. The piece was selected for its consistent tempo of 55-60 beats per minute (BPM) and stable average sound level of 60 decibels (dB). Music was played in the waiting room using a JBL Go3 speaker, with audio transmitted wirelessly via Bluetooth from a Huawei Nova 5T smartphone (Huawei, China). To maintain consistency, the speaker volume was calibrated each morning using the Sound Meter application (Google Play Store), ensuring the sound level remained at approximately 60 dB-comparable to normal conversational volume. Inside the OR, music was played directly from a computer with an attached speaker, and the same calibration method was applied. This volume level was chosen to avoid disrupting the surgeon's focus while allowing clear verbal communication between operating theatre staff and the participant. After listening to music for at least 15 minutes, participants were called into the OR according to their sequence. The same music continued to play in the OR for the music group until the end of the procedure.

Upon entering the OR, baseline samples of salivary alpha-amylase (sAA_before), BP (BP₁), and HR (HR₁) were measured. Salivary alpha-amylase (sAA) was assessed using the Cocoro Meter (Nipro Inc., Japan). Participants in the control group underwent the same procedure without background music.

All participants, regardless of group allocation, received standard IVI in accordance with clinical practice. The injections were performed under topical anaesthesia using five drops of proparacaine hydrochloride 0.5%, administered at least five minutes before the procedure. The periocular skin was cleaned with 10% povidone-iodine, while the conjunctiva and fornices were irrigated with 5% povidone-iodine and left for three minutes. The eye was then draped, and an eyelid speculum was applied. IVIs were performed under sterile conditions using a 30-gauge needle inserted 3.5-4.0 millimetres from the limbus.

During IVI, additional measurements of BP (BP₂) and HR (HR₂) were taken at the third minute. A second sAA measurement (sAA_after) was also obtained. Participants' pain levels were assessed using the Visual Analogue Scale for Pain (VAS-P).

Since approximately 30 patients were scheduled for IVI on any given day, their sequence of IVI was categorised for statistical analysis as early (8:00-10:00 a.m.), middle (10:00 a.m.-12:00 p.m.), and late (12:00-2:00 p.m.).

The duration of the procedure, type of anti-vascular endothelial growth factor (anti-VEGF) used, participant sequence, ocular diagnosis, number of prior IVIs, and history of ocular surgery were all documented. Each participant was recruited only once for the study, and no follow-up was required.

ELIGIBILITY:
Inclusion Criteria:

* patients who were Malaysia citizens aged 18 and above scheduled for elective intravitreal injection of anti-vascular endothelial growth factor (VEGF),
* capable of providing informed consent prior to trial participation.

Exclusion Criteria:

* patients with cognitive impairment precluding informed consent,
* patients with hearing impairment,
* patients with underlying psychological or psychiatric disorder,
* patients with prior salivary gland or facial surgery that could alter saliva secretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Salivary alpha amylase level | Periprocedural
  Salivary alpha amylase level was measured in kilo units per liter (KUnits/L). It was one of the objective biomarkers to measure anxiety in this study. It was measured right before injection and the 3rd minute after injection.
Blood pressure | Periprocedural
  Blood pressure was one of the anxiety markers measured in this study. It was measured in mmHg (millimetres of mercury) using an automated sphygmomanometer that had been calibrated in accordance with the manufacturer's recommended schedule prior to the commencement of the study.
  Several measurements were taken: on arrival at the day-care centre, on arrival at the operating room, and at the third minute after the intravitreal injection.
Heart rate | Periprocedural
  Heart rate was one of the anxiety markers measured in this study. It was measured in beats per minute (bpm) using an automated sphygmomanometer that had been calibrated in accordance with the manufacturer's recommended schedule prior to the commencement of the study.
  Several measurements were taken: on arrival at the day-care centre, on arrival at the operating room, and at the third minute after the intravitreal injection.
Perceived pain | Periprocedural
  Pain score measured using visual analogue scale for pain upon completion of intravitreal injection.
  It is presented as a 100 mm horizontal line, with numerical values ranging from 0 (no pain) to 10 (worst imaginable pain) distributed evenly along the line. Patients are instructed to indicate their current pain level by marking a point on the scale that best represents their experience. This scale is adapted from the Ministry of Health Malaysia's pain assessment guidelines and is routinely utilised in clinical settings in the country.

CONTACTS AND LOCATIONS:
Overall Officials: Ng Yu Siang Doctor, Principal Investigator — Universiti Malaya
Locations (1):
- Daycare Center, University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
to protect the confidentiality of the data of study participants

REFERENCES:
- [Background] Sugimoto K, Kanai A, Shoji N. The effectiveness of the Uchida-Kraepelin test for psychological stress: an analysis of plasma and salivary stress substances. Biopsychosoc Med. 2009 Apr 3;3:5. doi: 10.1186/1751-0759-3-5. PMID 19341484
- [Background] Chatterton RT Jr, Vogelsong KM, Lu YC, Ellman AB, Hudgens GA. Salivary alpha-amylase as a measure of endogenous adrenergic activity. Clin Physiol. 1996 Jul;16(4):433-48. doi: 10.1111/j.1475-097x.1996.tb00731.x. PMID 8842578
- [Background] Takai N, Yamaguchi M, Aragaki T, Eto K, Uchihashi K, Nishikawa Y. Effect of psychological stress on the salivary cortisol and amylase levels in healthy young adults. Arch Oral Biol. 2004 Dec;49(12):963-8. doi: 10.1016/j.archoralbio.2004.06.007. PMID 15485637
- [Background] Iizuka N, Awano S, Ansai T. Salivary alpha-amylase activity and stress in Japan air self-defense force cargo pilots involved in Iraq reconstruction. Am J Hum Biol. 2012 Jul-Aug;24(4):468-72. doi: 10.1002/ajhb.22247. Epub 2012 Feb 18. PMID 22344628
- [Background] Noto Y, Sato T, Kudo M, Kurata K, Hirota K. The relationship between salivary biomarkers and state-trait anxiety inventory score under mental arithmetic stress: a pilot study. Anesth Analg. 2005 Dec;101(6):1873-1876. doi: 10.1213/01.ANE.0000184196.60838.8D. PMID 16301277
- [Background] Anderson LC, Garrett JR, Johnson DA, Kauffman DL, Keller PJ, Thulin A. Influence of circulating catecholamines on protein secretion into rat parotid saliva during parasympathetic stimulation. J Physiol. 1984 Jul;352:163-71. doi: 10.1113/jphysiol.1984.sp015284. PMID 6205147
- [Background] Skov Olsen P, Kirkegaard P, Rasmussen T, Magid E, Poulsen SS, Nexo E. Adrenergic effects on secretion of amylase from the rat salivary glands. Digestion. 1988;41(1):34-8. doi: 10.1159/000199729. PMID 2462520
- [Background] Batzri S, Selinger Z. Enzyme secretion mediated by the epinephrine -receptor in rat parotid slices. Factors governing efficiency of the process. J Biol Chem. 1973 Jan 10;248(1):356-60. No abstract available. PMID 4348211
- [Background] Bellocchio L, Soria-Gomez E, Quarta C, Metna-Laurent M, Cardinal P, Binder E, Cannich A, Delamarre A, Haring M, Martin-Fontecha M, Vega D, Leste-Lasserre T, Bartsch D, Monory K, Lutz B, Chaouloff F, Pagotto U, Guzman M, Cota D, Marsicano G. Activation of the sympathetic nervous system mediates hypophagic and anxiety-like effects of CB(1) receptor blockade. Proc Natl Acad Sci U S A. 2013 Mar 19;110(12):4786-91. doi: 10.1073/pnas.1218573110. Epub 2013 Mar 4. PMID 23487769
- [Background] Hız M, Ciğerci Y, Doğan M. The effects of the music intervention on anxiety, pain, vital signs, and patient satisfaction in intravitreal injection: a randomized controlled study. Anatolian Clinic the Journal of Medical Sciences. 2022;27(2):150-61.
- [Background] Chan JC, Chan LP, Yeung CP, Tang TW, O YM, Lam WC. Effect of Music on Patient Experience during Intravitreal Injection. J Ophthalmol. 2020 Jul 30;2020:9120235. doi: 10.1155/2020/9120235. eCollection 2020. PMID 32802492
- [Background] Brosh K, Roditi E, Wasser LM, Aryan A, Hanhart J, Potter MJ. Effect of Music Selection on Anxiety Level during Intravitreal Injections for Individuals of Varying Cultures. Ophthalmic Epidemiol. 2022 Oct;29(5):582-587. doi: 10.1080/09286586.2021.1955390. Epub 2021 Jul 22. PMID 34293998
- [Background] Chen X, Seth RK, Rao VS, Huang JJ, Adelman RA. Effects of music therapy on intravitreal injections: a randomized clinical trial. J Ocul Pharmacol Ther. 2012 Aug;28(4):414-9. doi: 10.1089/jop.2011.0257. Epub 2012 Apr 16. PMID 22506884
- [Background] Richard-Lalonde M, Gelinas C, Boitor M, Gosselin E, Feeley N, Cossette S, Chlan LL. The Effect of Music on Pain in the Adult Intensive Care Unit: A Systematic Review of Randomized Controlled Trials. J Pain Symptom Manage. 2020 Jun;59(6):1304-1319.e6. doi: 10.1016/j.jpainsymman.2019.12.359. Epub 2019 Dec 24. PMID 31881291
- [Background] Beasley R. Pre-procedural education on anxiety levels during intravitreal injections. International Journal of Ophthalmic Practice. 2011;2(1):20-7.
- [Background] Jeong K, Kim J, Kim J, Hwang J. Relationship between Pain and Injection Site during Intravitreal Injection. Journal of the Korean Ophthalmological Society. 2016;57:930.
- [Background] Segal O, Segal-Trivitz Y, Nemet AY, Cohen P, Geffen N, Mimouni M. Anxiety levels and perceived pain intensity during intravitreal injections. Acta Ophthalmol. 2016 Mar;94(2):203-4. doi: 10.1111/aos.12802. Epub 2015 Jul 28. No abstract available. PMID 26215781
- [Background] Rifkin L, Schaal S. Factors affecting patients' pain intensity during in office intravitreal injection procedure. Retina. 2012 Apr;32(4):696-700. doi: 10.1097/IAE.0b013e3182252ad3. PMID 22082694